CLINICAL TRIAL: NCT04244513
Title: Deep Brain Stimulation Treatment for Chorea in Huntington's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Zhang Jianguo, Director of functional neurosurgery in Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2019-092-03
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Huntington Disease; Deep Brain Stimulation
Keywords: Deep brain stimulation; Chorea; Huntington Disease
MeSH Terms: conditions — Huntington Disease; Chorea | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups, of which the first group will be routinely activated after surgery and then stimulated for 6 months. The second group of patients will be re-launched 3 months after surgery, continued stimulation for 3 months, and then entered the open study. Patient data will be collected before surgery, 3 months after surgery, and 6 months after surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study adopts a blind design. One day before the first programming, the grouper and the programmer will release the cover independently. Only the grouper and the programmer will know the group information of each patient, in which the programmer does not communicate with the patient about the programming parameters. After each programming, the results are uniformly placed in the programmer to keep the others (patients, neurologists) blind about grouping and parameters. The evaluation will be finished by neurologists and video records of the patient's motor assessment. Neurologists do not participate in the surgical treatment and programmer. The statistical team is independent of other researchers. When performing statistical analysis, only the group information is known, the programming parameters corresponding to the group are blinded. The Medtronic company only provides equipment support and does not participate in any clinical research process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HD-DBS (Experimental): This group will be routinely activated after surgery and then stimulated for 6 months.
  Interventions: Device: Deep brain stimulation
- HD-sham-DBS (Sham Comparator): This group of patients will be re-launched 3 months after surgery, continued stimulation for 3 months
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — the HD-DBS arm will be routinely activated after surgery and then stimulated for 6 months(6 months stimulation). The HD-shamDBS arm will be re-launched 3 months after surgery, continued stimulation for 3 months(3 months stimulation), and then entered the open study.

SUMMARY:
1. Evaluating therapeutic effects of globus pallidus internus (GPi) deep brain stimulation (DBS) on Huntington's disease (HD) patients with chorea；
2. Explore the relationship between brain network conditions and DBS efficacy in HD patients
3. Explore the effect of different programmed parameters on the treatment of patients with DBS

DETAILED DESCRIPTION:
1. Evaluating therapeutic effects of GPi-DBS on HD patients with chorea: Clinical data of patients at different treatment time points will be collected, using different clinical assessments. The clinical case report form for HD-DBS is consistent with Enroll HD project and the case report form is attached in the appendix. The main purpose is to determine the efficiency of DBS treatment for HD with chorea by comparing the patients' status before and after surgery.

Primary endpoints: Changes in chorea score of UHDRS, changes in total motor score (UHDRS).

Secondary endpoints: changes in cognition will be assessed by stroop interference test, stroop word reading test, stroop colour naming test, trail making test, symbol digit modality test and mini-mental state examination(MMSE); changes in anxiety assessed by Hamilton Anxiety Scale(HAMA); changes in depression assessed by Hamilton depression scale(HAMD) and Beck Depression Inventory (BDI); changes in the frequency and severity of neuropsychiatric symptoms assessed by the Problem Behaviours Assessment for HD and changes in quality-of-life assessed by UHDRS functional assessment and UHDRS total functional capacity assessment.

2 Explore the relationship between brain network conditions and DBS efficacy in HD patients The electrophysiological signals during the operation of HD patients will be collected and analyzed, and compared with the postoperative disease conditions, to determine the relationship between the patient's EEG activity and the mechanism of disease development, disease progression, and treatment effect.

3. Explore the effect of different programmed parameters on the treatment of patients with DBS After the HD patient is turned on, the patient is programmed to adjust the program control parameters of different patients during adjustment, and the effects of different program control parameters on the patient, tolerance, and related side effects are clarified.

ELIGIBILITY:
Inclusion Criteria:

1. Huntington's Disease disgnosis by gene
2. Predominant chorea
3. UHDRS score ≥30
4. Mini-Mental State Examination (MMSE) score meets the education level
5. No plan to change medication within 12 months after randomization
6. Agree to enroll into the clinical trial

Exclusion Criteria:

1. Chorea caused by other diseases
2. Concurrently or previously had other neurological disorders
3. Severe psychiatric disease
4. Unstable condition or severe heart, lung, liver, kidney, or hematopoietic diseases
5. Have a history of cancer unless it has been cured or does not require treatment for the next 5 years
6. Contraindications to an MRI scan
7. Acute psychiatric symptomatology in the last 2 months including suicide ideation, angry or aggressive behaviour, and hallucinations

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale（UHDRS）-total score difference | 3 months postoperatively compared between groups
  Difference between groups in the UHDRS total score at 3 months postoperative；from 0 to 124 points; the higher scores mean a worse outcome
Unified Huntington's Disease Rating Scale（UHDRS）-total score difference | 6 months postoperatively compared with baseline
  Difference in the UHDRS total score at 6 months postoperative compared with baseline

SECONDARY OUTCOMES:
UHDRS-Chorea subscore difference | 6 months postoperatively compared with baseline
  Difference in the UHDRS chorea subscore at 6 months postoperative compared with baseline
Mental Behavior Rating Scale difference | 6 months postoperatively compared with baseline
  the total score of MMSE at 6 months postoperative compared with baseline
Mental Behavior Rating Scale difference | 6 months postoperatively compared with baseline
  the total score of BDI at 6 months postoperative compared with baseline
EuroQol five dimensions questionnaire (EQ-5D) difference | 6 months postoperatively compared with baseline
  the total score of EQ-5D at 6 months postoperative compared with baseline
Neuroimage | preoperative, 3 months and 6 months postoperative
  MRI
electrophysiology | 3 to 5 days postoperative
  EEG and Local field potential (LFP) of GPi and GPe in patients with Huntington's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, Ph.D, Study Chair — Beijing Tiantan Hospital
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No